CLINICAL TRIAL: NCT05573204
Title: Comparative Study Evaluating the Outcome of Obeticholic Acid Versus Vitamin E in Patients with Non-alcoholic Steatohepatitis Without Cirrhosis
Brief Title: Comparative Study Between Obeticholic Acid Versus Vitamin E in Patients with Non-alcoholic Steatohepatitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hadier Mohammed El-Sheikh, Assistant lecturer of clinical pharmacy- Clinical pharmacy department- Faculty of pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34512/2/21
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: NAFLD, non alcoholic fatty liver, fatty liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — obeticholic acid; Vitamin E

STUDY DESIGN:
Intervention Model Description: This study is randomized controlled, parallel and prospective 6-months duration study. Accepted patients will be randomized into 2 groups as the following:
  * Group 1 (Obeticholic acid group): 30 patients will receive 10 mg/day OCA for 6 months.
  * Group 2 (Control group): 30 patients will receive Vitamin E 400 mg twice daily for 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 obeticholic acid group (Active Comparator): 28 non alcoholic steatohepatitis patients receiving obeticholic acid 10 mg once daily for 6 months duration
  Interventions: Drug: Obeticholic Acid Oral Tablet
- Group 2 vitamin E group (Active Comparator): 31 non alcoholic steatohepatitis patients receiving vitamin E 400 mg twice daily for 6 months duration
  Interventions: Drug: Vit E

INTERVENTIONS:
Drug: Obeticholic Acid Oral Tablet — Obeticholic acid used as 10 mg tablet once daily for 6 months
  Other Names: Nashiliv 10 mg
  Arms: Group 1 obeticholic acid group
Drug: Vit E — Vitamin E used as 400 mg soft gelatin capsules twice daily for 6 months
  Other Names: Vitamin E 400 mg
  Arms: Group 2 vitamin E group

SUMMARY:
This study aims at evaluating and comparing the protective outcomes of using Obeticholic acid versus Vitamin E in NASH patients without cirrhosis. The intervention is 6-months duration and the study will assess the efficacy of either drug as fibrosis improvement (≥ 1 stage) with no worsening of NASH or NASH resolution with no worsening of fibrosis with the study considered successful if either 1ry end point is met. . Also, assessment of biochemical markers related to steatosis, inflammation, oxidative stress, insulin resistance and liver fibrosis will be done.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is defined as the accumulation of excessive fat in the liver in the setting of no significant alcohol consumption and the absence of any secondary cause. NAFLD has reached epidemic proportions and currently affects 20-40% of the general population. In recent years, along with the increasing trend of obesity and type 2 diabetes, NAFLD has become one of the most common chronic liver diseases worldwide. The spectrum of the disease ranges from simple steatosis to hepatocellular injury with inflammatory infiltration characterized as nonalcoholic steatohepatitis (NASH) that may eventually progress to liver fibrosis, cirrhosis and hepatocellular carcinoma. Despite significant disease burden and mortality associated mainly with advanced disease, i.e., NASH and fibrosis, there is currently no approved medication for NASH, therefore, lifestyle modifications remain the mainstay of treatment. What is the pathogenesis of NAFLD? Although the proposal of "two hits" involving insulin resistance (IR) and oxidative stress has been well accepted, the mechanism of NAFLD was thought very complex and still remained unclearly.

Farnesoid X receptor (FXR) is a nuclear hormone receptor, which is expressed in various organs and tissues, mainly in the liver, intestine, kidney, and adrenal cortex. It is a ligand activated transcription factor, with bile acid being the natural ligand to these receptors. These receptors are involved in regulating various metabolic pathways such as bile acid, cholesterol, and lipid and glucose metabolism. The expression of FXR is reduced in the liver of NASH patients, and various FXR knockout animal models exhibit hepatic steatosis, bile acid accumulation, hyperlipidaemia, hyperglycaemia and fibrosis. Importantly, these conditions are improved by increasing FXR expression, indicating that the FXR agonist could be an effective therapeutic option for NASH patients.

FXR activation significantly impacts lipid synthesis, mainly by decreasing the expression of the sterol regulatory element binding protein 1c (SREBP-1c) and its enzymes which are the main regulator in lipogenesis. In addition, FXR activation increases the clearance of LDL, very low density lipoprotein (VLDL) and chylomicrons by activation of lipoprotein lipase. Furthermore, FXR activation results in the induction of the peroxisome proliferator activated-α receptor which increases fatty acid oxidation. Also it increases the secretion of Fibroblast Growth Factor-21 (FGF-21) which decreases lipogenesis by inhibition of SREBP-1c.

Obeticholic acid (OCA) is a semisynthetic derivative of the chenodeoxycholic acid. OCA was originally described as a selective and potent FXR ligand. OCA is currently approved for treatment of primary biliary cholangitis. Currently, OCA is investigated for its potential role in the treatment of NASH. Phase II and III ongoing trials have shown that OCA might attenuate the severity of liver fibrosis in patients with NASH. In summary, OCA has been the first-in-class of FXR ligands advanced to a clinical stage, highlighting the potential benefits linked to FXR-targeted therapies.

It is acknowledged that vitamin E is the major lipid-soluble chain-breaking antioxidant found in the human body. In addition to its anti-oxidative properties, molecules of vitamin E family exert anti-atherogenic and anti-inflammatory activities. According to American Association for the Study of Liver Diseases (AASLD) and National Institute for Health and Care Excellence (NICE) guidelines, vitamin E is approved at a dose of 800 IU/day in adults with biopsy-proven NASH.

Therefore, This study aims at evaluating and comparing the protective outcomes of using Obeticholic acid versus Vitamin E in NASH patients without cirrhosis.

The primary endpoint of this 6-months study would be fibrosis improvement (≥ 1 stage) with no worsening of NASH or NASH resolution with no worsening of fibrosis with the study considered successful if either 1ry end point is met.

The secondary endpoint of this study is improvement of biochemical markers related to steatosis, inflammation, oxidative stress, insulin resistance and liver fibrosis.

Study Population:

* This study is conducted on 60 patients diagnosed with NASH according to the study protocol.
* Patients has been recruited from Tropical Medicine and Infectious Diseases Department, Tanta University Hospital, Tanta, Egypt.
* The study was approved by the Research Ethics Committee of Tanta University.
* All patients have provided signed written informed consent and agreed to comply with the study protocol.
* All data of the patients will be private and confidential.
* Any unexpected risks appeared during the course of the research was cleared to the patients and the ethical committee on time.

This study is randomized controlled, parallel and prospective 6-months duration study. Accepted patients was randomized into 2 groups as the following:

* Group 1 (Obeticholic acid group): 30 patients will receive 10 mg/day OCA for 6 months.
* Group 2 (Control group): 30 patients will receive Vitamin E 400 mg twice daily for 6 months.

Any side effects will be reported and graded according to common terminology criteria for adverse events version 5.00 (CTCAE). Any potential drug interactions between administered drugs is monitored for each patient and corrective actions is taken.

Statistical Analysis

* All data will be represented as mean ± slandered deviation (SD).
* Unpaired Student's t-test will be used to compare data between the two groups.
* Paired Student's t-test will be used to compare data within the same group before and after treatment with the studied medications.
* Chi-square test will be used for statistical analysis of nominal data.
* The statistical analysis will be carried out using Statistical Package for the Social Sciences (SPSS) statistical package version 27.0 (December 2020), IBM (International Business Machines) corporation software group, USA.
* The level of significance will be set at P< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥18 years.
* All patients are diagnosed to have fatty liver grading 1, 2 or 3 on abdominal ultrasound with Hepatic steatosis index > 36 to be considered as a NAFLD patient.
* Confirmed diagnosis of NASH using at least three of the following non-invasive tests:
* HAIR score
* Fibroscan detecting steatosis with F0-3 fibrosis stage
* Cytokeratin-18 >240 U/L
* Mild to moderate elevation of serum aminotransferases (>2 but <5 times upper normal limit)

Exclusion Criteria:

* Current or history of significant alcohol consumption.
* Use of drugs historically associated with nonalcoholic fatty liver disease (NAFLD) (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, and other known hepatotoxins).
* Prior or planned bariatric surgery.
* Uncontrolled diabetes defined as Hemoglobin A1c 9.5% or higher.
* Evidence of other forms of chronic liver disease as Hepatitis B, Hepatitis C, Wilson's disease, Alpha-1-antitrypsin(A1AT) deficiency, Hemochromatosis, drug-induced liver disease.
* Serum creatinine of 2.0 mg/dL or greater.
* Pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the trial and breast feeding.
* Use of other drugs known to have possible positive effects on steatosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-10-25 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline fibrosis stage at 6 months; fibrosis improvement (≥ 1 stage), with no worsening of steatosis, detected by fibroscan device | 6 months
  Patients will undergo fibroscan testing prior to the initiation of the intervention and after 6 months of receiving the drug therapy to detect fibrosis improvement
Change from baseline steatosis stage at 6 months with no worsening of fibrosis detected by Fibroscan device | 6 months
  Patients will undergo fibroscan testing prior to the initiation of the intervention and after 6 months of receiving the drug therapy to detect steatosis improvement

SECONDARY OUTCOMES:
Change in serum level of fibroblast growth factor-21(FGF-21) | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate fibroblast growth factor-21(FGF-21)
Change in serum level of cytokeratin-18 (CK-18) | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate cytokeratin-18 (CK-18)
Change in serum level of Liver enzymes; Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alk. Phosphatase (ALP) and Gamma-glutamyl transferase (GGT)
Change in HAIR SCORE | 6 MONTHS
  HAIR score decrease or increase
change in BMI | 6 months
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Hadier m. El-sheikh, Principal Investigator — Department of Clinical pharmacy, Faculty of Pharmacy, Tanta university
Locations (1):
- Department of Tropical Medicine and Infectious Diseases, Faculty of Medicine,Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Venetsanaki V, Karabouta Z, Polyzos SA. Farnesoid X nuclear receptor agonists for the treatment of nonalcoholic steatohepatitis. Eur J Pharmacol. 2019 Nov 15;863:172661. doi: 10.1016/j.ejphar.2019.172661. Epub 2019 Sep 16. PMID 31536725
- [Background] Yang ZX, Shen W, Sun H. Effects of nuclear receptor FXR on the regulation of liver lipid metabolism in patients with non-alcoholic fatty liver disease. Hepatol Int. 2010 Aug 12;4(4):741-8. doi: 10.1007/s12072-010-9202-6. PMID 21286345
- [Background] Fuchs M. Non-alcoholic Fatty liver disease: the bile Acid-activated farnesoid x receptor as an emerging treatment target. J Lipids. 2012;2012:934396. doi: 10.1155/2012/934396. Epub 2011 Dec 7. PMID 22187656
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- See also: Obeticholic action; all you need to know — http://go.drugbank.com/drugs/DB05990